CLINICAL TRIAL: NCT06825806
Title: Femoral Artery Doppler Indices as an Emerging Predictor of Spinal Anesthesia-induced Hypotension in Elective Cesarean Section: A Prospective Observational Study
Brief Title: Doppler Indices to Predict Spinal Hypotension During Cesarean Section
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, lecturer of anesthesia and critical care, Cairo University
Other Study IDs: Doppler and spinal hypotension
Record Dates: First submitted 2025-02-08; First posted 2025-02-13 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-02

CONDITIONS: Spinal Hypotension; Doppler
Keywords: Spinal hypotension; Cesarean section; femoral Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Femoral artery Doppler — Right common femoral artery will be examined before and after spinal anesthesia to evaluate pulsatility index, resisitive index, and waveform morphology

SUMMARY:
Spinal anesthesia is safe and advisable anesthetic during cesarean section, despite that spinal induced hypotension is a common associated problem. Therefore early recognition of these critical events should take high priority to avoid serious consequences. in this regards several parameters were available to detect spinal hypotension but non is satisfactory till now. Researchers of this study aimed to evaluated the diagnostic accuracy of femoral artery Doppler to predict hypotension

ELIGIBILITY:
Inclusion Criteria:

* ASA II
* singleton pregnancy
* full term

Exclusion Criteria:

* vascular disease
* contraindication to spinal anesthesia
* inability to obtain adequate Doppler

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women undergoing cesarean section
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Accuracy of the change in pulsatility index to predict spinal hypotension | baseline and immediately after spinal anesthesia

SECONDARY OUTCOMES:
accuracy of change in waveform morphology to predict spinal hypotension | baseline and immediately after spinal anesthesia
baseline shock index to predict hypotension | baseline
baseline PI to predict spinal hypotension | baseline
baseline RI to predict hypotension | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Helmy, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Data regarding this research will be available from the corresponding author upon reasonable request

REFERENCES:
- [Background] Yu C, Gu J, Liao Z, Feng S. Prediction of spinal anesthesia-induced hypotension during elective cesarean section: a systematic review of prospective observational studies. Int J Obstet Anesth. 2021 Aug;47:103175. doi: 10.1016/j.ijoa.2021.103175. Epub 2021 May 1. PMID 34034957
- [Background] Adolf Helmy M, Mansour M, Magdy Milad L, Mohammed Aboelregal E, Magdy Youssef M. Change in femoral artery pulsatility index as a novel predictor of post-spinal anesthesia hypotension in adult patients undergoing infra-umbilical surgeries: A prospective observational study. Anaesth Crit Care Pain Med. 2025 Apr;44(2):101482. doi: 10.1016/j.accpm.2025.101482. Epub 2025 Jan 21. No abstract available. PMID 39848332
- [Background] Kinsella SM, Carvalho B, Dyer RA, Fernando R, McDonnell N, Mercier FJ, Palanisamy A, Sia ATH, Van de Velde M, Vercueil A; Consensus Statement Collaborators. International consensus statement on the management of hypotension with vasopressors during caesarean section under spinal anaesthesia. Anaesthesia. 2018 Jan;73(1):71-92. doi: 10.1111/anae.14080. Epub 2017 Nov 1. No abstract available. PMID 29090733
- [Background] Kim ES, Sharma AM, Scissons R, Dawson D, Eberhardt RT, Gerhard-Herman M, Hughes JP, Knight S, Marie Kupinski A, Mahe G, Neumyer M, Poe P, Shugart R, Wennberg P, Williams DM, Zierler RE. Interpretation of peripheral arterial and venous Doppler waveforms: A consensus statement from the Society for Vascular Medicine and Society for Vascular Ultrasound. Vasc Med. 2020 Oct;25(5):484-506. doi: 10.1177/1358863X20937665. Epub 2020 Jul 15. PMID 32667274
- See also: Related Info — https://doi.org/10.1016/j.accpm.2025.101482